CLINICAL TRIAL: NCT01212211
Title: Hyponatremia in the Elderly: Benefit From a Change in Drug Therapy?
Acronym: NATRIPHAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-A00778-31
Record Dates: First submitted 2010-09-10; First posted 2010-09-30 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Sodium level; Falls; Gait; elderly
MeSH Terms: conditions — Hyponatremia | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- change in drug therapy (Experimental): Change in drug therapy with the help of the opinion of pharmacologists : the physician would review the drug treatment of ten residents in coordination with the opinion of pharmacologists
  Interventions: Other: change in drug therapy
- reference (No Intervention): drug treatment of ten patients will remain unchanged during the three months of inclusion

INTERVENTIONS:
Other: change in drug therapy — Change in drug therapy with the help of the opinion of pharmacologists : the physician would review the drug treatment of ten residents in coordination with the opinion of pharmacologists
  Arms: change in drug therapy

SUMMARY:
Mild hyponatremia is the commonest electrolyte imbalance in the older population. Recently, association between hyponatremia and bone fractures in the ambulatory elderly has been shown.

Mild chronic hyponatremia is causing falls and lead to hospitalisation because of attention deficit.

Symptoms related to hyponatremia can be very subtle and difficult to detect clinically. Twenty elderly patients, retirement homes residents, with serum sodium < 135mEq/L will be included. They will be randomised. The physician will review the drug treatment of ten patients in coordination with the opinion of pharmacologists. Drug treatment for ten other patients wil remained unchanged during the three months of inclusion.

Useful elements of the medical records of patients randomized to the experimental arm will be forwarded to the Pharmacovigilance Regional Center for opinion pharmacologist. The notice, subject to the attention of physician of retirement homes, give rise to a therapeutic approach towards the patient. It will be followed by weekly monitoring of serum sodium for 4 weeks to evaluate the impact of the intervention. Thus, the effectiveness of medical intervention will be evaluated by an objective biological criteria: serum sodium in the fourth week. Secondary endpoints will evaluate the duration of normalization of serum sodium and check the interest of correcting hyponatremia to improve postural capacities and eventually reduce the number of falls in the medium term (three months).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 65 years Resident of dependent elderly
* Plasma sodium <135 mmol / l less than a week, confirming earlier hyponatremia within a week to three month agreement given after patient information

Exclusion Criteria:

* Venous system does not allow sampling - Patient not taking medication-Dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the benefit of a change of drug therapy following a review pharmacologist on the increase in serum sodium in elderly | Fourth week
  Normalization serum sodium between S0 and S4 (4 weeks after medical intervention)

SECONDARY OUTCOMES:
Normalization of serum sodium-Evaluate the impact on the deficit postural S4-Evaluate the impact on the occurrence of falls | three months
  Changes in serum sodium weekly S1, S2, S3 - Evolution of the score evaluation of postural control: the Timed Up and Go test (TUG) between therapeutic intervention and S4-comparison of the number of falls between the period three months before and three months after surgery Medical Decision to three months whether to maintain the drug therapy changed

CONTACTS AND LOCATIONS:
Overall Officials: Blandine De la Gastine, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Centre Hospitalier Carentan, Carentan, France